CLINICAL TRIAL: NCT02073422
Title: Fractional Flow Reserve Versus Angiographically Guided Management to Optimise Outcomes in Unstable Coronary Syndromes - a 3.0 Tesla Stress Perfusion MRI Sub-Study (FAMOUS-NSTEMI MRI)
Brief Title: FAMOUS-NSTEMI MRI Sub-Study
Status: Completed | Type: Observational
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: University of Glasgow (Other); British Heart Foundation (Other); NHS Lanarkshire (Other Government); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Colin Berry, Professor of Cardiology and Imaging, NHS National Waiting Times Centre Board
Other Study IDs: NRS-11-CA56, PG/11/55/28999; PG/11/55/28999 (Other Grant/Funding Number: British Heart Foundation PG/11/55/28999)
Record Dates: First submitted 2014-02-19; First posted 2014-02-27 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: NonST Elevation Myocardial Infarction
Keywords: Magnetic resonance imaging; Myocardial stress perfusion magnetic resonance imaging; Fractional flow reserve; Relaxometry; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-ST elevation myocardial infarction: Natural history study of non-ST elevation myocardial infarction and coronary physiology
  Interventions: Device: Fractional flow reserve; Other: Magnetic resonance imaging

INTERVENTIONS:
Device: Fractional flow reserve — Guidewire-based index of coronary artery stenosis severity measured when coronary microvascular resistance is minimised by administration of a vasodilator drug.
  Other Names: FFR
Other: Magnetic resonance imaging — Cardiac magnetic resonance imaging at 3.0 Tesla, including perfusion MRI at rest and during pharmacological stress with intravenous adenosine (140-210 ug/kg/min).
  Other Names: MRI

SUMMARY:
BACKGROUND: Non-ST-segment elevation myocardial infarction (NSTEMI) is the commonest type of acute coronary syndrome (ACS) and has a poor long-term prognosis. Guidewire-based coronary pressure measurement of the myocardial fractional flow reserve (FFR) is validated for measuring the severity of a coronary lesion narrowing in patients with stable angina. FFR measurement in patients with a recent ACS has theoretical limitations and is not fully validated.

AIM: To prospectively assess heart muscle blood flow and injury with guide-wire based methods at the time of the clinically-indicated angiogram and compare these results with those from a stress perfusion MRI scan in medically-stabilised NSTEMI..

HYPOTHESIS: 1) FFR measured invasively will correspond closely with findings from stress perfusion MRI, 2) MRI will provide clinically-relevant information on heart muscle injury, function and salvage, 3) Guidewire-derived measurements of coronary microvascular function will be associated with the MRI findings.

DESIGN: The MRI study will be performed in patients who give informed consent in the FAMOUS-NSTEMI clinical trial (NCT registration 01764334). All of the clinical data for these participants will be available to link with the MRI results.

DETAILED DESCRIPTION:
BACKGROUND: Non-ST elevation myocardial infarction (NSTEMI) is the commonest type of acute coronary syndrome (ACS) and has a poor long-term prognosis. Guidewire-based coronary pressure measurement of the myocardial fractional flow reserve (FFR) is a prognostically-validated invasive method for measuring coronary lesion severity in patients with stable coronary artery disease. FFR measurement in patients with unstable coronary disease has theoretical limitations and is not fully validated in NSTEMI.

AIM: To prospectively evaluate ischaemia and infarction with adenosine stress perfusion cardiac MRI in medically-stabilised NSTEMI patients in whom FFR has been measured.

METHODS: In the FAMOUS-NSTEMI clinical trial (NCT registration 01764334), medically-stabilised patients with recent NSTEMI will have lesion-level ischaemia measured with FFR in all coronary artery stenoses amenable to revascularisation, as clinically appropriate.

Consecutive study participants will be invited to have an adenosine (140 µg/kg/min) stress 3.0 Tesla cardiac MRI scan to assess myocardial perfusion on up to three occasions: 1) before coronary angiography, 2) within 10 days post coronary angiography and finally, 3) 6 months after hospital admission. MRI will also assess myocardial pathophysiology including ischaemia, oedema, haemorrhage and infarct scar. MRI will provide the reference dataset. Guidewire-derived parameters were obtained and assessed blind to the MRI results.

The primary outcome is the correspondence between the presence or absence of an inducible-myocardial perfusion defect and FFR ≤ or > 0.80 in the MRI scans at baseline or post-angiography. Secondary outcomes include the correlation between measures of infarct severity as revealed by MRI (infarct size, myocardial salvage, microvascular obstruction, myocardial haemorrhage, myocardial strain) and invasive measures of coronary function (1) coronary collateral supply (fractional coronary collateral supply), (2) microcirculatory resistance (index of microvascular resistance), and (3) vasodilator capacity (resistive reserve ratio).

The project was funded by the British Heart Foundation and Chief Scientist Office. The pressure wires were provided through a restricted grant from St Jude Medical. The funders of the study have no involvement in the study design, analysis, interpretation, or presentation of the results.

VALUE: This study will provide clinically important information on the relationships between coronary artery and microcirculatory function measured invasively and ischaemia and MI pathologies, as revealed by non-invasively by MRI.

ELIGIBILITY:
Inclusion Criteria:

* (1) Participation in the FAMOUS NSTEMI clinical trial (NCT registration 01764334); (2) age >18 years; (3) written informed consent.

Exclusion Criteria:

* 1) Contra-indications to MRI including metallic devices and severe kidney disease (i.e. an estimated glomerular filtration rate <30 ml/min/1.73 m2).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medically stabilised patients with recent non-ST elevation myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2014-06-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Correspondence between FFR and myocardial perfusion revealed by adenosine stress perfusion MRI. | MRI at baseline
  FFR is a guidewire based measurement of lesion-level flow limitation during hyperaemia. An MRI perfusion defect is classified as significant according to the presence of ischaemia in 2 segments of a 32 segment model i.e: > 60 degrees in either the basal or the mid-ventricular slices or > 90 degrees in the apical slice or any transmural defect or two adjacent slices. FFR and MRI will be correlated in corresponding coronary artery territories based on coronary anatomy. The analysis is for diagnostic accuracy of FFR vs. myocardial perfusion as assessed by MRI in temporally associated assessments at baseline.

SECONDARY OUTCOMES:
Myocardial Infarction | Baseline MRI scan
  Presence and extent (% left ventricular volume) of infarction, as revealed by late gadolinium contrast enhancement.
Myocardial area-at-risk | Baseline MRI scan
  The myocardial ischaemic area-at-risk revealed by non-contrast MRI methods (T1 mapping, T2 mapping, T2-weighted MRI).
Myocardial salvage | Baseline and follow-up MRI (average 12 months)
  Myocardial salvage is estimated by subtraction of infarct size from the initial area-at-risk. Salvage may be estimated at baseline with initial infarct size or at follow-up (final infarct size).
Myocardial salvage index | Baseline and follow-up MRI (average 12 months)
  Myocardial salvage index is estimated by indexing infarct size to the initial area-at-risk. Salvage may be estimated at baseline with initial infarct size or at follow-up with final infarct size.
Left ventricular ejection fraction | Baseline and follow-up MRI (average 12 months)
  Left ventricular ejection fraction (LVEF) is an index of left ventricular systolic function, and a surrogate outcome measure of treatment efficacy and patient outcome.
Culprit artery assignment | Baseline MRI scan
  Magnetic resonance imaging of myocardial ischaemic injury with non-contrast MRI methods should theoretically identify the culprit artery in patients with a recent non-ST elevation myocardial infarction. The MRI methods to be used in this study include T1 mapping (MOLLI, Siemens Healthcare), T2 mapping (bSSFP, Siemens Healthcare) and T2-STIR (dark blood oedema MRI). The diagnostic accuracy of these three methods will be compared using a combination of clinical parameters (ECG, coronary angiogram, invasive adjunctive diagnostic methods, contrast enhanced MRI) which together represent the reference dataset for culprit artery assignment in individual patients.
Microvascular obstruction | Baseline MRI scan
  Microvascular obstruction revealed by MRI is due to a failure of gadolinium contrast to diffuse into the infarct zone because of extrinsic compression (e.g. oedema) and intrinsic obstruction (e.g. microvascular thrombosis).
Myocardial haemorrhage | Baseline MRI
  Myocardial haemorrhage is a consequence of vascular damage and is related to the duration of ischaemia, infarct severity and coronary reperfusion. Transverse (T2) and T2* magnetisation are destroyed by the paramagnetic effects of deoxyhaemoglobin. Signal loss in T2*-weighted images have high positive predictive accuracy for myocardial haemorrhage. T2 and T2* mapping methods, and STIR (dark blood MRI) will be used to assess the incidence of haemorrhage.
Regional myocardial strain | Baseline and follow-up MRI (average 12 months)
  Myocardial strain is an intrinsic property of myocardial contractility. Left ventricular (LV) thickening and inward LV motion (which is how LVEF is calculated) are passive phenomena secondary to active circumferential shortening and sources of artefact (such as through plane motion) can misrepresent actual LV contractility. Strain-encoded cardiac MRI with DENSE will be used to assess regional strain in the left ventricle, segmented according to the American Heart Association model. The mid-ventricular level will be a particular region of interest.
Adenosine response | Baseline
  FFR and perfusion MRI require systemic vasodilatation. In this study, systemic hyperaemia is induced by administration of intravenous adenosine (140 ug/kg/min - 210 ug/kg/min). The patient response (symptoms, haemodynamics, MRI) will be assessed prospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, MB ChB BSc FRCP FACC, Principal Investigator — University of Glasgow
Locations (1):
- BHF Glasgow Cardiovascular Research Centre, Glasgow, Strathclyde, United Kingdom

REFERENCES:
- [Background] Berry C, Layland J, Sood A, Curzen NP, Balachandran KP, Das R, Junejo S, Henderson RA, Briggs AH, Ford I, Oldroyd KG. Fractional flow reserve versus angiography in guiding management to optimize outcomes in non-ST-elevation myocardial infarction (FAMOUS-NSTEMI): rationale and design of a randomized controlled clinical trial. Am Heart J. 2013 Oct;166(4):662-668.e3. doi: 10.1016/j.ahj.2013.07.011. Epub 2013 Aug 27. PMID 24093845
- [Background] Layland J, Rauhalammi S, Watkins S, Ahmed N, McClure J, Lee MM, Carrick D, O'Donnell A, Sood A, Petrie MC, May VT, Eteiba H, Lindsay M, McEntegart M, Oldroyd KG, Radjenovic A, Berry C. Assessment of Fractional Flow Reserve in Patients With Recent Non-ST-Segment-Elevation Myocardial Infarction: Comparative Study With 3-T Stress Perfusion Cardiac Magnetic Resonance Imaging. Circ Cardiovasc Interv. 2015 Aug;8(8):e002207. doi: 10.1161/CIRCINTERVENTIONS.114.002207. PMID 26253733
- [Background] Layland J, Rauhalammi S, Lee MM, Ahmed N, Carberry J, Teng Yue May V, Watkins S, McComb C, Mangion K, McClure JD, Carrick D, O'Donnell A, Sood A, McEntegart M, Oldroyd KG, Radjenovic A, Berry C. Diagnostic Accuracy of 3.0-T Magnetic Resonance T1 and T2 Mapping and T2-Weighted Dark-Blood Imaging for the Infarct-Related Coronary Artery in Non-ST-Segment Elevation Myocardial Infarction. J Am Heart Assoc. 2017 Mar 31;6(4):e004759. doi: 10.1161/JAHA.116.004759. PMID 28364045